CLINICAL TRIAL: NCT02971358
Title: Safety and Early Efficacy of Radical Prostatectomy for Newly Diagnosed Very High Risk Locally Advanced and Oligometastatic Prostate Cancer - a Prospective Single Center Phase I/II Study
Brief Title: Safety and Early Efficacy of Radical Prostatectomy for Newly Diagnosed Very High Risk Locally Advanced and Oligometastatic Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Bernhard Grubmüller, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1461/2016
Record Dates: First submitted 2016-11-20; First posted 2016-11-22 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced and Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radical prostatectomy arm (Experimental): In this arm the investigators will include patients with locally advanced or metastatic prostate cancer, who will undergo cytoreductive radical prostatectomy with extended lymph node dissection.
  Interventions: Procedure: Radical prostatectomy

INTERVENTIONS:
Procedure: Radical prostatectomy — Standard radical prostatectomy with extended lymph node dissection is performed.

SUMMARY:
Prostate cancer is the most common non-skin cancer diagnosed among men and the second leading cause of male cancer deaths in the United States. In 2013, it is estimated that 29,270 men have died from prostate cancer. Although radiation and surgery are quite effective for localized disease, there is no effective cure for men who present with metastatic prostate cancer as the 5-year relative survival rate is only 28%.

Currently, androgen deprivation therapy (ADT) via medical or surgical castration is the standard first-line therapy in men with metastatic disease but castration-recurrent prostate cancer (CRPC) eventually emerges with a median time of 18-24 months. Once CRPC develops, secondary hormonal manipulation, chemotherapy, and immunotherapy are marginally effective.

Given the dismal prognosis of metastatic prostate cancer, new ideas and novel approaches must be explored to improve the clinical outcome. In this regard, recently emerging data suggest that local tumor control may enhance the effectiveness of subsequent systemic therapies. Therefore, in this proposal, the investigators have designed a Phase I/II study in which they will prospectively evaluate the safety and feasibility of cytoreductive prostatectomy in men with newly diagnosed mPCa.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Very high risk PCA (PSA ≥ 20 oder Gleason Score ≥ 8 oder ≥ cT3) and/or oligometastasierte PCA (T any N positive M any, oder T any N any M positive)
* ≤5 bone metastasis
* ≤75 years
* Ability for informed consent
* Clinically no infiltration into the rectum or pelvic wall
* Clinically no visceral metastasis
* Male, >18 Jahre
* Fit for surgery
* ECOG Performance Status 0 oder 1

Exclusion Criteria:

* Male, < 18 Jahre
* > 5 bone metastasis
* > 75 years
* No ability for informed consent
* Clinically infiltration into the rectum or pelvic wall
* Not fit for surgery
* Clinically visceral metastasis

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The rate of perioperative complications within 90 days after surgery (Clavien-Dindo-classification) | 90

SECONDARY OUTCOMES:
Time to start androgen deprivation therapy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided